CLINICAL TRIAL: NCT03282851
Title: Randomized, Double-Blind, Parallel-Group, Single-Dose Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, Tolerability and Immunogenicity of MSB11456, US-licensed Actemra® and EU-approved RoActemra® in Healthy Adult Subjects
Brief Title: Pharmacokinetics/Pharmacodynamics (PK/PD) Equivalence Study of MSB11456
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MS200740-0001
Record Dates: First submitted 2017-08-30; First posted 2017-09-14 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: MSB11456; Actemra®; RoActemra®
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MSB11456 (Experimental)
  Interventions: Drug: MSB11456
- US-licensed Actemra (Active Comparator)
  Interventions: Drug: US-licensed Actemra
- EU-approved RoActemra (Active Comparator)
  Interventions: Drug: EU-approved RoActemra

INTERVENTIONS:
Drug: MSB11456 — Subjects will receive a single injection of MSB11456 on Day 1.
  Arms: MSB11456
Drug: US-licensed Actemra — Subjects will receive a single injection of US-licensed actemra on Day 1.
  Arms: US-licensed Actemra
Drug: EU-approved RoActemra — Subjects will receive a single injection of EU-approved RoActemra on Day 1.
  Arms: EU-approved RoActemra

SUMMARY:
This study aims to compare the PK/PD of a single injection of investigational Medicinal Product (IMP) MSB11456, US licensed Actemra and EU approved RoActemra in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 55 years of age, with a body mass index (BMI) between 18 and 29.9 kilogram per meter square (kg/m^2).
* Subjects who are on adequate contraception as defined in the protocol and are willing and able to comply with the scheduled study visits, Investigational medicinal product (IMP) administration, safety laboratory tests, and all other study procedures.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Subjects with history and/or current presence of clinically significant atopic allergy (for example, asthma including childhood asthma, urticaria, angio-edema, eczematous dermatitis).
* Subjects with hypersensitivity or allergic reactions, including known or suspected clinically relevant drug hypersensitivity to any components of the IMP formulations, comparable drugs, or to latex.
* Subjects who have active or latent tuberculosis as indicated by a positive QuantiFERON®-Tuberculosis (TB) Gold test or a history of tuberculosis, lifetime history of invasive systemic fungal infections (for example, histoplasmosis) or other opportunistic infections, including recurrent or chronic local fungal infections, frequent (more than 3 per year requiring treatment) chronic or recurrent infections, having previously been treated with tocilizumab or taken a recombinant monoclonal antibody.
* Subjects who have received a live vaccine within 12 weeks before enrolling in this study or planning for any such vaccination during the study or within 4 months after IMP administration.
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 696 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Serum Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-t) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48
Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48
Maximum Observed Serum Concentration (Cmax) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48

SECONDARY OUTCOMES:
Area Under Curve From Tme Zero to 72 Hours After Dosing (AUC 0-72) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48
Percentage of Area Under Curve From Zero to Infinity (AUC0-∞) Obtained by Extrapolation (AUC extra%) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48
Time To Reach Maximum Serum Concentration (tmax) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48
Time to Last Observed Serum Concentration (tlast) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48
Apparent Terminal Rate Constant (λz) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48
Apparent Terminal Half-life (t½) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48
Apparent Total Body Clearance of Drug from Serum Following Subcutaneous Administration (CL/F) of MSB11456, US-licensed Actemra, and EU-approved RoActemra | Up to Day 48
Safety Profile as Assessed by Incidence of Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), Injection Site Reactions, Laboratory Variables, Vital Signs and Electrocardiogram (ECG) Measurements | Up to Day 48
Immunogenicity as Assessed by Incidence of Antidrug Antibodies (ADAs), Neutralizing Antibodies (NABs) | Up to Day 48

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Fresenius Kabi SwissBioSim GmbH
Locations (2):
- New Zealand (2):
  - Research site, Auckland
  - Research site, Christchurch